CLINICAL TRIAL: NCT01239342
Title: A Randomized Phase 2 Study of MK-2206 in Comparison With Everolimus in Refractory Renal Cell Carcinoma
Brief Title: Akt Inhibitor MK2206 or Everolimus in Treating Patients With Refractory Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-02270; NCI-2010-02270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 8727; MDA-2010-0247; CDR0000688457; 2010-0247; 8727 (Other: M D Anderson Cancer Center); 8727 (Other: CTEP); N01CM00038 (NIH); N01CM00039 (NIH); N01CM62202 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Kidney Carcinoma; Recurrent Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — MK 2206; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Akt inhibitor MK2206) (Experimental): Patients receive Akt inhibitor MK2206 PO on days 1, 8, 15, and 22. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who are progression free after 1 year may receive a 12 week study drug supply of Akt inhibitor MK2206.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis
- Arm II (everolimus) (Experimental): Patients receive everolimus PO QD on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
  Arms: Arm I (Akt inhibitor MK2206)
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
  Arms: Arm II (everolimus)
Other: Laboratory Biomarker Analysis — Optional correlative studies

SUMMARY:
This randomized phase II trial studies the side effects and how well Akt inhibitor MK2206 or everolimus works in treating patients with kidney cancer that does not respond to treatment. Akt inhibitor MK2206 and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Everolimus may also stop the growth of kidney cancer by blocking blood flow to the tumor. It is not yet known whether Akt inhibitor MK2206 or everolimus is more effective in treating kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess progression free survival (PFS) of vascular endothelial growth factor (VEGF) therapy refractory renal cell carcinoma (RCC) patients who receive either MK-2206 (Akt inhibitor MK-2206) or everolimus.

II. To assess safety of MK-2206 in patients with VEGF therapy refractory RCC.

SECONDARY OBJECTIVES:

I. To assess overall response rate (ORR) and overall survival (OS). (Clinical) II. To assess time to treatment failure (TTF). (Clinical) III. To determine whether baseline AKT activation is predictive for clinical benefit after treatment with MK-2206 or everolimus. (Pre-clinical/exploratory) IV. To determine whether circulating cytokines and angiogenic factors predict for clinical benefit after treatment with MK-2206 or everolimus. (Pre-clinical/exploratory) V. To assess impact of karyotype on outcome in patients treated with MK-2206 or everolimus. (Pre-clinical/exploratory)

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive Akt inhibitor MK2206 orally (PO) on days 1, 8, 15, and 22. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who are progression free after 1 year may receive a 12 week study drug supply of Akt inhibitor MK2206.

ARM II: Patients receive everolimus PO once daily (QD) on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or unresectable RCC; all histologies are permitted; patient should have undergone nephrectomy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients must have received, and progressed on an anti-VEGF therapy, including bevacizumab, sorafenib, sunitinib or pazopanib
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN; therapeutic anticoagulation with warfarin is allowed if target INR =< 3 on a stable dose of warfarin or on a stable dose of low molecular weight (LMW) heparin for > 2 weeks at time of randomization
* Women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 8 weeks after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Serum pregnancy test in female patients of childbearing potential must be negative within 24 hours of enrolling on this study

Exclusion Criteria:

* Patients who received oral tyrosine-kinase inhibitors (TKIs) (sorafenib, sunitinib, or pazopanib) within 2 weeks prior to entering the study, radiotherapy, immunotherapy or chemotherapy within 4 weeks prior to entering the study, bevacizumab within 4 weeks prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier (recovered to =< grade 1)
* Patients may not be receiving any other investigational agents; patients may not have received an mammalian target of rapamycin (mTOR) inhibitor
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or other agents used in the study
* Patients receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP4503A4) are ineligible
* Patient should have a hemoglobin A1C value of < 8%; preclinical studies demonstrated the potential of MK-2206 for induction of hyperglycemia in all preclinical species tested; studies also demonstrate a risk of hyperglycemia, hyperlipidemia and hypertriglyceridemia associated with everolimus therapy; patients with diabetes or in risk for hyperglycemia, hyperlipidemia and/or hypertriglyceridemia should not be excluded from trials with MK-2206 or everolimus, but the patient should be well controlled on oral agents (recent [i.e. within 3 months] hemoglobin [Hb]A1C =< 7.0) before the patient enters the trial
* Baseline corrected Fridericia QT interval (QTcF) > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MK-2206 or everolimus
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Individuals who are diagnosed with an intercurrent cancer are excluded, with the exception of non-melanoma skin cancers, and other cancers where curative treatment was completed at least two years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-01-27 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, Principal Investigator — M.D. Anderson Cancer Center
Locations (8):
- United States (8):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 27, 2011 to January 9, 2013. All recruitment done in medical clinic settings.
Groups:
- MK2206: Akt inhibitor MK2206 200 mg orally once weekly, courses repeat every 4 weeks.
- Everolimus: Everolimus 10 mg orally once daily, courses repeat every 4 weeks.
Period: Overall Study
Arm/Group | MK2206 | Everolimus
Started | 29 | 14
Completed | 26 | 8
Not Completed | 3 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Reason Unknown | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK2206 | Everolimus | Total
Number analyzed (Participants) | 29 | 14 | 43
Age, Continuous [Median (Full Range); unit: years] | 59 [43 to 83] | 63.5 [48 to 84] | 62 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 21 | 14 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 28 | 9 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 26 | 14 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 14 | 43

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS) in Months
Description: PFS defined as Time interval between date of treatment and date of disease progression, date of death or last follow-up date, whichever occurs first. Progression defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a nontarget lesion, or the appearance of new lesions.
Time Frame: Time interval between date of treatment and date of disease progression, date of death or last follow-up date, whichever occurs first, assessed up to 5 years
Population: One participant in each group left study before restaging therefore are excluded from response outcome analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MK2206 | Everolimus
Number analyzed (Participants) | 28 | 13
Months | 3.68 [1.77 to 5.75] | 5.98 [5.03 to NA] — Trial met futility criteria at the planned interim analysis therefore full confidence interval was not estimable.

2. Secondary Outcome: Clinical Benefit Defined as Number of Participants With Complete Response (CR) + Partial Response (PR) + Stable Disease (SD)
Description: Clinical benefit defined as participants' with CR+PR+SD assessed using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Repeat radiologic studies to evaluate disease progression or response (in accordance with restaging of disease) every 8 weeks. Complete Response (CR): Disappearance all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): >30% decrease in sum diameters of target lesions, reference baseline sum diameters. Progressive Disease (PD): >20% increase in sum diameters of target lesions, reference smallest sum on study (includes baseline sum if is smallest on study). In addition to relative increase of 20%, sum must demonstrate absolute increase >5 mm. (Note: appearance 1/+ new lesions considered progressions). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum diameters.
Time Frame: Up to 5 years
Population: One participant in each group left study before restaging therefore are excluded from outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MK2206 | Everolimus
Number analyzed (Participants) | 28 | 13
Participants
  Complete Response | 1 | 0
  Partial Response | 3 | 0
  Stable Disease | 11 | 11
  Progressive Disease | 13 | 2

3. Secondary Outcome: Summary of Selected Toxicities Grade 3 or Greater Toxicity Based on the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Adverse Events (AEs) list of reported events with associated intervention agent in a uniform presentation of events. The method of Thall, Simon and Estey (1995, 1996) was used to collect study participants' safety data summarized by treatment arm, category, severity and relevance. Comprehensive listing of AEs collected on study can be found in Adverse Event section separated by severity, Serious and Other AEs and represented by treatment arm, organ system-category within defined severity.
Time Frame: Up to 5 years
Measure: Number; unit: Toxicities
Arm/Group | MK2206 | Everolimus
Number analyzed (Participants) | 29 | 14
Toxicities
  Hyperglycemia | 7 | 1
  Hypertriglyceridemia | 1 | 1
  Hyperuricemia | 2 | 0
  Lymphocyte count decreased | 2 | 1
  Mucositis oral | 1 | 0
  Rash maculo-papular | 8 | 0
  Pruritus | 1 | 0
  Proteinuria | 1 | 0
  Pancreatitis | 1 | 0
  Lipase increased | 1 | 0
  Generalized muscle weakness | 1 | 0
  Dyspnea | 1 | 0
  Dehydration | 2 | 0

4. Secondary Outcome: Overall Response Rate (ORR) Defined as Complete Response (CR) + Partial Response (PR)
Description: Response for CR + PR defined by RECIST version 1.1. Repeat radiologic studies to evaluate disease progression or response (in accordance with restaging of disease) every 8 weeks. Complete Response (CR): Disappearance all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): >30% decrease in sum diameters of target lesions, reference baseline sum diameters. Progressive Disease (PD): >20% increase in sum diameters of target lesions, reference smallest sum on study (includes baseline sum if is smallest on study). In addition to relative increase of 20%, sum must demonstrate absolute increase >5 mm. (Note: appearance 1/+ new lesions considered progressions). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum diameters.
Time Frame: Up to 5 years
Population: One participant in each group left study before restaging therefore are excluded from response outcome analysis.
Measure: Number; unit: percentage of participants
Arm/Group | MK2206 | Everolimus
Number analyzed (Participants) | 28 | 13
percentage of participants | 14.3 | 0

5. Secondary Outcome: Median Overall Survival (OS) in Months
Description: Overall survival reported in months as time interval between the date of treatment and the date of death or last follow-up.
Time Frame: Time interval between the date of treatment and the date of death or last follow-up, assessed up to 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | MK2206 | Everolimus
Number analyzed (Participants) | 29 | 14
Months | 23.5 [10.7 to 37.4] | 15.7 [6.5 to NA] — "NA" as this value is not estimable due to the small sample size which generated a very wide confidence interval.

6. Secondary Outcome: Time to Failure (TTF)
Description: TTF defined as Time interval between the date of treatment and the date of disease progression, date of death, date of treatment discontinuation due to severe toxicity or last follow-up date.
Time Frame: Time interval between the date of treatment and the date of disease progression, date of death, date of treatment discontinuation due to severe toxicity or last follow-up date, assessed up to 5 years
Population: No participants analyzed. Data not collected.
Arm/Group | MK2206 | Everolimus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected through each 28 day course, and reporting for events that occur within 30 Days of the last dose of the investigational agent.
Arm/Group | MK2206 | Everolimus
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/14
Serious Adverse Events (participants affected / at risk) | 7/29 | 2/14
Other Adverse Events (participants affected / at risk) | 29/29 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK2206 (N=29) | Everolimus (N=14)
Death NOS (General disorders) | 4 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK2206 (N=29) | Everolimus (N=14)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 3
Activated partial thromboplastin time prolonged (Investigations) | 18 | 3
Alanine aminotransferase increased (Investigations) | 4 | 1
Alkaline phosphatase increased (Investigations) | 11 | 7
Allergic reaction (Immune system disorders) | 2 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4
Anemia (Blood and lymphatic system disorders) | 24 | 11
Anorexia (Metabolism and nutrition disorders) | 5 | 3
Anxiety (Psychiatric disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 4
Ataxia (Nervous system disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 5
Bloating (Gastrointestinal disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac disorders - (Other), specify (Cardiac disorders) | 2 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Chills (General disorders) | 0 | 1
Cholesterol high (Investigations) | 17 | 12
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Creatinine increased (Investigations) | 25 | 10
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Depression (Psychiatric disorders) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 11 | 7
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dry eye (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1
Dysesthesia (Gastrointestinal disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Ear pain (Ear and labyrinth disorders) | 2 | 0
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 10 | 7
Endocrine disorders - (Other), specify (Endocrine disorders) | 11 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye disorders - (Other), specify (Eye disorders) | 2 | 0
Fatigue (General disorders) | 24 | 12
Fever (General disorders) | 4 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flatulence (General disorders) | 1 | 0
Gait disturbance (Musculoskeletal and connective tissue disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - (Other), specify (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 3
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hemoglobinuria (Renal and urinary disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 28 | 10
Hyperkalemia (Metabolism and nutrition disorders) | 10 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1
Hyperthyroidism (Endocrine disorders) | 8 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 20 | 12
Hyperuricemia (Metabolism and nutrition disorders) | 14 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 1
Hyponatremia (Metabolism and nutrition disorders) | 10 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 1
Hypotension (Vascular disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1
Infections and infestations - (Other), specify (Infections and infestations) | 3 | 5
Injury, poisoning and procedural complications - (Other) (Injury, poisoning and procedural complications) | 0 | 1
INR increased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Investigations - (Other) (Investigations) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lipase increased (Investigations) | 1 | 0
Localized edema (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Lymphocyte count decreased (Investigations) | 20 | 10
Mucositis oral (Gastrointestinal disorders) | 13 | 7
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Specify (Other) (Musculoskeletal and connective tissue disorders) | 2 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nervous system disorders - (Other), specify (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 2
Non-cardiac chest pain (General disorders) | 2 | 2
Pain (General disorders) | 10 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 1
Palpitations (Cardiac disorders) | 1 | 0
Papulopustular rash (Infections and infestations) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Platelet count decreased (Investigations) | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 15 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 24 | 6
Rash pustular (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - (Other), specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1
Serum amylase increased (Investigations) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Surgical and medical procedures - (Other), specify (Surgical and medical procedures) | 2 | 2
Thromboembolic event (Vascular disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 2
Watering eyes (Eye disorders) | 6 | 3
Weight loss (General disorders) | 4 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
White blood cell decreased (Investigations) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT01239342/Prot_SAP_000.pdf